CLINICAL TRIAL: NCT07137975
Title: Assessment of Bone Volume Using Patient Specific Autogenous Bone Plug Versus Particulate Autogenous Bone for Unilateral Alveolar Ridge Reconstruction: A Randomized Clinical Trail
Brief Title: Assessment of Bone Volume Using Patient Specific Autogenous Bone Plug Versus Particulate Autogenous Bone for Unilateral Alveolar Ridge Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Raed, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS3-3-14
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Alveolar Cleft Grafting
Keywords: Alveolar Cleft; Cleft; Grafting; Ridge Augmentation; 3D defect

STUDY DESIGN:
Intervention Model Description: Preoperative assessment of the alveolar defect began with intraoral examination to check a proper transverse relationship between the maxillary segments and the presence of a normal upper arch form.
  After the decision on alveolar bone grafting, Radiologic data from the cleft area will be required. Standard protocol is to take a high resolution CT scan of the patient's skull or at least the whole maxilla. Using the DICOM data acquired from the cleft area the bony defect will be segmented with specific software, in our daily routine blender for dental is used. The same program could be used to design the rough shape of the nasoalveolar graft, and this image could be exported in STL (standard tessellation language) format. and once the desired form is aquired, the final step is to construct a mold. For this purpose, the open-source software Blender (Blender Foundation, Amsterdam, and The Netherlands) will be used. After preoperative planning, the designed mold will be printed using polyam
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenous bone plug (Active Comparator)
  Interventions: Other: autogenous bone plug
- control (Experimental)
  Interventions: Other: regular autogenous bone grafting

INTERVENTIONS:
Other: autogenous bone plug — Preoperative assessment of the alveolar defect began with intraoral examination to check a proper transverse relationship between the maxillary segments and the presence of a normal upper arch form.
  After the decision on alveolar bone grafting, Radiologic data from the cleft area will be required. Standard protocol is to take a high resolution CT scan of the patient's skull or at least the whole maxilla. Using the DICOM data acquired from the cleft area the bony defect will be segmented with specific software, in our daily routine blender for dental is used. The same program could be used to design the rough shape of the nasoalveolar graft, and this image could be exported in STL (standard tessellation language) format. and once the desired form is aquired, the final step is to construct a mold. For this purpose, the open-source software Blender (Blender Foundation, Amsterdam, and The Netherlands) will be used. After preoperative planning, the designed mold will be printed using polyam
  Arms: autogenous bone plug
Other: regular autogenous bone grafting — Gold standard grafting of alveolar cleft
  Arms: control

SUMMARY:
Most common complications that arise from alveolar cleft repair surgeries are; failure of graft integration, wound dehiscence, scar tissue formation, infections, bone exposure and oral-nasal fistula formation.

Alveolar cleft patients have compromised soft tissue which increase the chance of graft exposure.

To Augment the alveolar defect in three-dimensions, accurate assessment of alveolar cleft is essential, virtual surgical planning can be combined with 3D printing to re-create the defect virtually. Based of virtually created defect a patient specific mold can be designed. Printed mold will be used as a medium for adding particulate autogenous graft mixed with fibrin glue creating a plug with the precise shape of the alveolar cleft, the fibrin glue will assist in forming the plug as well as acting as a scaffold for migrating fibroblasts as well as a hemostatic barrier, stimulates mesenchymal cell, induces and promotes angiogenesis, and also initiates early osteogenesis.

DETAILED DESCRIPTION:
-The aim of this study is to describe an auxiliary surgical techniques in alveolar cleft reconstruction and evaluate volume of the bone.

Research question:

Does the use of patient specific autogenous plug yield better 3D volume than conventional autogenous graft.

Statement of the problem:

Cleft patients need a precise treatment regimen, which makes the treatment challenging. Multidisciplinary approach is required and collaboration of multiple specialties is needed; OMFS, orthodontists, plastic surgeons, speech therapist and pedodontists. One of the most crucial steps in treatment of cleft patients is the repair of the alveolar defect to achieve stability of the arch, provide room for canine and lateral incisor to erupt, maintain periodontal health of adjacent teeth, restore continuity of piriform rim, support the ala of the nose to allow for better facial appearance, closure of oronasal fistula to decrease chance URT infections and allow for better hygiene and speech., It is essential to understand and evaluate the geometry and size of the defect, to avoid improper grafting of the defect, enhance the evaluation of the alveolar defect preoperatively, and the graft integration postoperatively and to allow precise repair of the alveolar defect. (Watted et al., 2020) (Stolarz et al.,2022) Each alveolar cleft has a unique shape in mesio-distally, antro-posteriorly, which creates a challenge to fill the defect in all dimensions. The precise assessment of the cleft geometry can be determined by computed tomography (CT), or cone- beam CT (CBCT) which allows simultaneous alveolar cleft assessment, planning and volume measurement.

4

Rationale for conducting the research:

Most common complications that arise from alveolar cleft repair surgeries are; failure of graft integration, wound dehiscence, scar tissue formation, infections, bone exposure and oral-nasal fistula formation.

Alveolar cleft patients have compromised soft tissue which increase the chance of graft exposure.

To Augment the alveolar defect in three-dimensions, accurate assessment of alveolar cleft is essential, virtual surgical planning can be combined with 3D printing to re-create the defect virtually. Based of virtually created defect a patient specific mold can be designed. Printed mold will be used as a medium for adding particulate autogenous graft mixed with fibrin glue creating a plug with the precise shape of the alveolar cleft, the fibrin glue will assist in forming the plug as well as acting as a scaffold for migrating fibroblasts as well as a hemostatic barrier, stimulates mesenchymal cell, induces and promotes angiogenesis, and also initiates early osteogenesis. (Kesztyűs et al., 2022)

ELIGIBILITY:
1. Inclusion criteria:

   * Patients with unilateral alveolar clefts who completed pre-operative expansion.
   * Patients with good oral hygiene.
   * Patients free from any medical condition that might compromise the healing process.
   * Both males and females will be included in trail.
   * Age range from 7 years to 12 years.
2. Exclusion criteria:

   * Unmotivated/uncooperative patients and/or parents.
   * Patients who previously underwent unsuccessful treatment trails.
   * Patients with insufficient ridge expansion.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage fill | 6 months

SECONDARY OUTCOMES:
bone density | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt